CLINICAL TRIAL: NCT06466174
Title: Determination of the Safety and Efficacy of Two Probiotic Strains in Adults With Mild to Moderate Gastrointestinal Discomfort
Brief Title: Determination of the Safety and Efficacy of Two Probiotic Strains
Acronym: CODECS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Merieux NutriSciences (China) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PCTB202108
Record Dates: First submitted 2024-05-16; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Gastrointestinal Dysfunction
Keywords: probiotic; gastrointestinal discomfort

STUDY DESIGN:
Intervention Model Description: Placebo crossover to probiotic A Probiotic A crossover to Placebo Placebo crossover to probiotic B Probiotic B crossover to Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo 1 to Probiotic A (Active Comparator): Sequence A1 (n=25): Placebo 1 administered daily for 42 days, followed by 21 days washout, then 1 x 10^9 colony forming units (CFU) of Probiotic A administered daily for 42 days
  Interventions: Dietary Supplement: Placebo 1 to Probiotic A
- Placebo 2 to Probiotic B (Active Comparator): Sequence B1 (n=25): Placebo 2 administered daily for 42 days, followed by 21 days washout and 42 days Probiotic formula: containing 1 x 10^9 CFU of Probiotic B administered daily
  Interventions: Dietary Supplement: Placebo 2 to Probiotic B
- Probiotic A to Placebo 1 (Active Comparator): Sequence A2 (n=25): 1 x 10^9 CFU of Probiotic A administered daily for 42 days, followed by 21 days washout, then Placebo 1 administered daily for 42 days
  Interventions: Dietary Supplement: Probiotic A to Placebo 1
- Probiotic B to Placebo 2 (Active Comparator): Sequence B2 (n=25): 1 x 10^9 CFU of Probiotic B administered daily for 42 days, followed by 21 days washout and 42 days Placebo 2 administered daily for 42 days
  Interventions: Dietary Supplement: Probiotic B to Placebo 2

INTERVENTIONS:
Dietary Supplement: Placebo 1 to Probiotic A — 42 day Crossover study design between Placebo 1 and Probiotic A (n = 25)
  Arms: Placebo 1 to Probiotic A
Dietary Supplement: Probiotic A to Placebo 1 — 42 day Crossover study design between Probiotic A and Placebo 1 (n = 25)
  Arms: Probiotic A to Placebo 1
Dietary Supplement: Placebo 2 to Probiotic B — 42 day Crossover study design between Placebo 2 and Probiotic B (n = 25)
  Arms: Placebo 2 to Probiotic B
Dietary Supplement: Probiotic B to Placebo 2 — 42 day Crossover study design between Probiotic B and Placebo 2 (n = 25)
  Arms: Probiotic B to Placebo 2

SUMMARY:
The goal of this study is to determine the safety and efficacy of two probiotic strains in adults with mild to moderate gastrointestinal discomfort. The main questions it aims to answer is whether 6-week administration of a probiotic can improve how the participant feels regarding their gut health. This is done by completing a weekly questionnaire and the results are compared between the 6 weeks the participants are on a placebo and the 6 weeks the participants are on the probiotic. Participants will also provide a blood sample, and stool sample at the start and end of each treatment. Similarly, the results from the blood samples and stool samples will be analysed to determine if there is any improvement in markers related to gut health.

DETAILED DESCRIPTION:
In this randomized, crossover, double-blind, prospective, placebo controlled study we aim to determine the safety and efficacy of two probiotic strains in adults with mild to moderate gastrointestinal discomfort. 100 healthy adults with subclinical mild to moderate gastrointestinal complaints (GSRS-IBS score 20-45 inclusive), 50 subjects per strain (test sequence). The GSRS-IBS (gastrointestinal symptom rating scale - irritable bowel syndrome) questionnaire ranges from 0-78 with a greater score indicating a higher occurrence of gastrointestinal symptoms. Safety: To evaluate adverse events that occur during the probiotic treatment period as compared to the placebo period. Incidence and duration of upper respiratory tract symptoms, urinary tract symptoms, gastrointestinal symptoms as primary outputs. Efficacy: To evaluate the effect of 6-week probiotic administration on gastrointestinal homeostasis using GSRS-IBS score as an index as compared to placebo. Following a screening period, participants will provide stool, urine (safety) and blood samples prior to commencing a 6 week course of either placebo or one of the probiotics. At this time participants will again provide blood and stool samples. Throughout the study participants will maintain a daily diary to note any unusual events and to report stool consistency using Bristol stool chart. The participants will also complete a once-weekly questionnaire (GSRS-IBS questionnaire) relating to gut health. There will then be a 3-week washout period where they will take no products. After these 3 weeks the participants will again provide a stool and blood samples, and as before maintain their daily diary and weekly questionnaire for 6 weeks while on the probiotic or placebo (they will have swapped at this point). After these 6 weeks the participants will again provide stool and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent form
2. Healthy adults aged 18-65 years
3. Subclinical mild to moderate gastrointestinal complaints (GSRS-IBS score 20-45 at baseline)

Exclusion Criteria:

1. Presence of a serious congenital anomaly or chronic medical condition that would contraindicate participation, including history of major gastrointestinal surgery, chronic gastrointestinal illness, abnormal intestinal anatomy or significant abdominal disorder
2. Severe chronic illnesses
3. Known immunodeficiency
4. Use of immunosuppressive agents (corticosteroids, methotrexate…)
5. Presence of severe immunodeficient family members as provided by subjects self-report
6. Pregnancy, 6 months postpartum period or current breastfeeding
7. Women of childbearing age planning pregnancy during the course of the study
8. Actively participating in another clinical study, having completed a clinical study in the past 60 days or being in the exclusion period of a previous clinical study
9. Not able to understand and comply with requirements of the study
10. Use of probiotics, prebiotics, postbiotics, antibiotics within 3 weeks of study commencement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in GSRS-IBS score | Baseline vs Week 6
  Change in the GSRS-IBS score while participants are on the treatment as compared with placebo. GSRS-IBS ranges from 0-78 with a greater score indicating a higher occurence of gastrointestinal symptoms

SECONDARY OUTCOMES:
Incidence of upper respiratory tract symptoms | Baseline vs Week 6
  Incidence of upper respiratory tract symptoms, as captured by incidence of upper respiratory tract as reported by clinician/PI
Duration of upper respiratory tract symptoms | Baseline vs Week 6
  Duration of upper respiratory tract symptoms, as captured by duration of upper respiratory tract as reported by clinician/PI
Incidence of urinary tract infections | Baseline vs Week 6
  Incidence of urinary tract infections, as captured by incidence of urinary tract infections as reported by clinician/PI
Duration of urinary tract infections | Baseline vs Week 6
  Duration of urinary tract infections, as captured by duration of urinary tract infections as reported by clinician/PI

OTHER OUTCOMES:
Change in Stool consistency | Baseline vs Week 6
  To evaluate the difference in stool consistency as determined by daily Bristol stool chart scale captured in daily diary. The Bristol stool chart ranges from 1-7, with 1,2 being hard and solid and 6,7 being loose and watery. This readout will be the change in stool consistency towards types 3,4 and 5
Questionnaire regarding general health | Baseline vs Week 6
  General health questionnaire regarding mood, sleep, energy, concentration and changes in appetite. This is based on a Likert scale ranging from 0 (no effect) to 7 (severe)
Changes in microbiome readouts | Baseline vs Week 6
  To determine if there are any changes in alpha and beta diversity in the microbiome using 16S rRNA sequencing ( a common methodology used in assessing microbiome readouts) between placebo and probiotic treatment.
Changes in blood immune biomarkers | Baseline vs Week 6
  To determine if there are any changes in biomarkers relating to immune markers including IL-6 (IL interleukin), IL-10, TNFalpha, IFNgamma in pg/mL serum.
Regularity of defecation | Baseline vs Week 6
  Regularity of defecation as captured by daily diary
Changes in serum short chain fatty acid levels | Baseline vs Week 6
  Changes in serum short chain fatty acids (SCFA's) including acetate, propionate and butyrate in micromol/L)
Changes in serum amino acids levels | Baseline vs Week 6
  Changes in serum amino acids levels including the essential amino acids histidine, isoleucine, leucine, lysine, methionine, phenylalanine, threonine, tryptophan, and valine; and the non-essential amino acids alanine, arginine, asparagine, aspartic acid, cysteine, glutamic acid, glutamine, glycine, proline, serine, and tyrosine in micromol/L

IPD SHARING:
Plan to Share IPD: No